CLINICAL TRIAL: NCT00577980
Title: Testosterone Replacement Therapy in Castration-Resistant Prostate Cancer
Brief Title: Testosterone in Castration-Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Zero accrual and failure to generate multicenter interest.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0316
Record Dates: First submitted 2007-12-17; First posted 2007-12-20 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Castration-Resistant Prostate Cancer; Testosterone Replacement Therapy; Testosterone; CRPC; TRT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone (Experimental): Testosterone 200 mg administered parenterally by intramuscular (IM) injection every 2 weeks
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Initial dose of Testosterone 200 mg IM administered followed by 200 mg - 400 mg every 2 weeks.

SUMMARY:
Primary Objective:

1. To assess the prostate-specific antigen (PSA)-response (50% decline) to Testosterone Replacement Therapy (TRT) in men with "intermediate and good-risk" Castration-Resistant Prostate Cancer (CRPC).

Secondary Objectives:

1. To assess the objective response and time-to-progression with TRT in CRPC.
2. To assess serial changes in quality of life with TRT in these CRPC subsets.
3. Translational: To study kinetics of circulating tumor cells with TRT and molecular correlates of response to TRT in CRPC.

DETAILED DESCRIPTION:
Generally, castration therapy has been used indefinitely for prostate cancer patients because some tumors seem to grow faster with testosterone present. Researchers want to study the effect of testosterone only in patients whose tumors have had a maximum response to castration therapy. Researchers want to find out if these patients' disease may be better controlled with testosterone replacement therapy.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded and there will be a review of all medicines you may be currently taking. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate). You will have blood drawn (about 4 teaspoons) and urine collected for routine tests. You will have a chest x-ray, an electrocardiogram (ECG--a test to measure the electrical activity of the heart), a bone scan, and a computed tomography (CT) scan of your abdomen and pelvis. If the study doctor thinks it is necessary, you may have an assessment of your mental status. For this assessment, you will be asked questions about your attention span, memory, and mood disturbances. It will take about 25 minutes to complete.

If you are found to be eligible to take part in this study, you will begin receiving testosterone enanthate replacement therapy every 2 weeks by an injection into a muscle.

Every 2 weeks, you will go to the clinic for your testosterone injection, and blood (about 2 teaspoons) will be drawn to check the testosterone level in your blood. This will help the study doctor learn what dose you will receive for the next 2 weeks. After your Week 8 visit, blood (about 2 teaspoons) will be drawn to check the testosterone level in your blood every 4 weeks for the rest of your time on this study.

At the Week 8 and 24 visits, you will have a physical exam, including measurement of your vital signs. You will be asked about any side effects you may be experiencing. Your disease status will be evaluated to learn its response to treatment. Blood (about 4 teaspoons) will be drawn for routine tests, and you will have repeat imaging scans (like the ones you had at your screening visit) to evaluate your disease. If the study doctor thinks that your mental status should be assessed again, you will have another assessment (at or around Week 24) like the one completed during your screening visit.

You may remain on this study indefinitely unless your disease gets worse or you experience any intolerable side effects.

If your participation ends on this study for any of the above reasons, you will have an end-of-study visit. During this visit, you will have blood drawn (about 4 teaspoons) for routine testing. You will be asked about any side effects you may be experiencing, and your disease response to treatment will be evaluated.

This is an investigational study. Testosterone enanthate is commercially available. Testosterone replacement therapy is not FDA approved for this disease, and in some cases, has been disallowed for use in prostate cancer. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a history of histologically or cytologically confirmed adenocarcinoma of the prostate.
* Patients must have had a history of a response to medical or surgical castration therapy for prostate cancer with a serum PSA nadir of </= 0.2 ng/ml and must not have had any known subsequent rise in serum PSA level of any magnitude above this nadir within the first 24 months of hormonal therapy. Nadir PSA value following hormonal therapy in combination with non-hormonal therapy such as radical prostatectomy, radiation therapy or chemotherapy do not count towards eligibility.
* Patients must have current evidence of progressive castration-resistant disease that is asymptomatic. Progressive disease is defined by a) radiological evidence of progression: any increase of > 25% in the products of diameters or 30% in maximum diameter of any measurable lesion; or appearance of an unequivocally new lesion OR b) two consecutive rises in serum PSA of any magnitude measured at least 2 weeks apart, to a level above 2 ng/ml.
* Patients must have a minimum serum PSA level of 1 ng/ml.
* Patients may have palpable disease or radiological evidence of metastatic disease but without the following high-risk features: lymphangitic lung disease on chest X-ray or CT scan; bilateral hydronephrosis related to prostate cancer, palpable disease in the prostate, known brain metastases or suspicion of impending spinal cord or nerve root compression.
* Patients must have a documented castrate level of testosterone (</= 50ng/ml). For patients who are medically castrated, luteinizing hormone releasing hormone analog will continue. The purpose is to simplify and harmonize exogenous testosterone therapeutics.
* Patients on anti-androgens should be discontinued from such therapy for at least 4 weeks (for bicalutamide for at least 6 weeks), prior to initiation of testosterone therapy and must have had documented progression of disease as in #3.
* Patients must satisfy the following laboratory criteria: serum total bilirubin < 2 * institutional upper limit of normal (ULN) and serum aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) </= 2.5 * institutional ULN.
* The Eastern Cooperative Oncology Group (ECOG) performance status 0-3.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Small cell or sarcomatoid prostate cancers are not eligible.
* No prior chemotherapy for CRPC.
* Patients may not be receiving any other investigational agents or hormonal therapy besides that specified in the study.
* Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infections defined as requiring IV antibiotics on day 1 of treatment or psychiatric illness/social situations that would limit compliance with study requirements.
* Unwilling or unable because of comorbid conditions to tolerate intramuscular injections of testosterone every 2 weeks.
* Overt psychosis, mental disability or otherwise incompetent to give informed consent or history of non-compliance.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Rate of Prostate Specific Antigen (PSA) - decline by 50% | Every 2 weeks, after Week 8 every 4 weeks till end of study
  Rate is the number of participants with PSA-response defined as PSA > or equal to 50%-decline in PSA from baseline value sustained for at least 4 weeks with be no evidence of progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org